CLINICAL TRIAL: NCT05686109
Title: Ancillary Study: Monitoring of Patients After Ambulatory Surgery by Biobeat® Devices: Pilot Feasibility Study
Brief Title: Substudy of MEET-OS (NCT04948632): Monitoring of Patients After Ambulatory Surgery by Biobeat® Devices
Acronym: BIOBEAT
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: HEC Montreal (Unknown)
Responsible Party: Sponsor
Other Study IDs: 22.220
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Surgery-Complications; Patient Satisfaction; Patient Compliance
Keywords: Monitoring device; Ambulatory surgery; Postoperative complications
MeSH Terms: conditions — Patient Satisfaction; Patient Compliance; Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monitoring device Biobeat®: Biobeat® non-invasive monitoring devices can be used in an out-of-hospital perioperative setting to observe patients' vital signs up to 5 days postoperatively.
  The Biobeat® portable adhesive device will be installed after the surgery, in the recovery room. All patients will be equipped with a portable single-use Biobeat® Bluetooth device that will be positioned at chest level and connected via Bluetooth to the patient's cell phone. These patches have been FDA approved since 2019 (new approval in 2022) for non-invasive (systolic, diastolic, and mean) blood pressure measurement without a cuff. The following other parameters will also be recorded: peripheral oxygen saturation, heart rate, respiratory rate and body temperature based on the analysis of the plethysmography wave. This data will be recorded as soon as the patches are installed.

SUMMARY:
The objective of this ancillary study of the MEET-OS study is to assess the technical feasibility of using Biobeat® monitoring devices after ambulatory surgery at high risk of complications.

The secondary objectives are to assess: i) the patient's experience and tolerance ii) the occurrence of clinical disturbances in the patients's home after ambulatory surgery with high risk of postoperative complications iii) to determine the impact of the data obtained with the monitoring devices on the clinical care decisions during postoperative follow-up.

DETAILED DESCRIPTION:
With increasingly complex surgeries and increasingly comorbid patients, ambulatory surgery are not always at low risk of postoperative complications. Among the new support tools available for monitoring patients remotely, devices for monitoring vital signs could be of interest to healthcare staff in charge of monitoring, more precisely when comorbid patients are involved or when interventions at high risk of complications are performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old undergoing elective outpatient surgery under general or regional anesthesia
* Internet access for the patient or their caregiver from home
* Written, oral and spoken comprehension of French
* Considered to be at high risk of postoperative complications, defined by one of the following two criteria: an ASA 3 score or an ASA score of 2 + surgery at intermediate or high risk according to the classification of Glance and al.

Exclusion Criteria:

* Patient's or caregiver's inability to learn and to use digital technologies
* Conversion of ambulatory to inpatient hospitalization on the day of surgery
* Patient's refusal
* Operation performed under regional or neuraxial anesthesia alone
* Trophic skin disorders contraindicating the installation of the Biobeat® monitoring device on the torso (deformation, irritation, infection, ulceration, etc.)
* Patient with pacemaker
* MRI or CT scheduled post-operatively
* Tattoo on the torso or refusal to shave the area where the Biobeat® monitoring device should be installed
* Pregnant or breastfeeding women
* Allergy to one of the technological components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent an ambulatory surgery considered at high-risk of postoperative complications at the CHUM, who have accepted to be enrolled in the main study MEET-OS with two groups of patients : a group benefiting from optimized support and follow-up using the LeoMed telecare platform (Group A) and a group benefiting from the current standard of care (Group B).
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with no loss of data for a period of 2 consecutive hours over the entire follow-up period. | From the installation of the monitoring device after the surgery up to 5 days postoperatively.

SECONDARY OUTCOMES:
Percentage of useful data available per day for the interpretation of vital signs during the first 5 days | From the installation of the monitoring device after the surgery up to 5 days postoperatively.
Percentage of patients with no data loss for 1, 4, 6, and 8 consecutive hours over the entire follow-up period. | From the installation of the monitoring device after the surgery up to 5 days postoperatively.
Percentage of patients with data loss of one hour or more preceding a postoperative event. | From the installation of the monitoring device after the surgery up to 5 days postoperatively.
  The postoperative event is defined as a call to the CHUM health info line.
Frequency of occurrences and the cumulative time of clinical disturbances | From the installation of the monitoring device after the surgery up to 5 days postoperatively.
  The occurrence of manufacturer alerts and the following clinical disturbances within 72 hours postoperatively will be evaluated: moderate postoperative arterial hypotension (defined by mean arterial pressure < 65 mmHg), severe arterial hypotension defined by MAP < 60 mmHg; moderate arterial hypertension defined by an MAP > 110mmHg; severe arterial hypertension defined by a MAP > 130mmHg; bradycardia defined by a heart rate < 40bpm; tachycardia defined by a heart rate > 100bpm; bradypnea defined by respiratory rate < 8/min; tachypnea defined by respiratory rate > 20/min; oxygen desaturation < 95%; oxygen desaturation < 90%; oxygen desaturation < 85%; hypothermia defined as body temperature < 36.0°C; hyperthermia defined as body temperature > 38.0°C.
Patient's experience | 7 days after the surgery
  A phone interview will be conducted to collect the patient's experience with a questionnaire derived from Breteler and al., which consist of 12 questions, adapted to the present study and focused on the experience of the patient and his caregiver, his tolerance and his satisfaction.
Percentage of appropriate and inappropriate clinical decision changes from the clinical intervention decided by the expert committee will be assessed. | Up to 60 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Florian Robin, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No